CLINICAL TRIAL: NCT02234258
Title: Cognitive Behavioral Social Skills Training for Youth at Risk of Psychosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: The Zucker Hillside Hospital (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jean Addington, PhD, Dr Jean Addington, University of Calgary
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: MH105178
Record Dates: First submitted 2014-09-03; First posted 2014-09-09 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: At Risk of Psychosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral social skills (Experimental): In Cognitive behavioral social skills training (CBSST), skills-based CBT is used to teach individuals how to correct inaccurate dysfunctional thoughts that interfere with goal-directed activities, including defeatist expectancies, low self-efficacy beliefs, and anomalous beliefs. SST focuses on behaviorally-based instruction of interpersonal social skills, utilizing role-modeling, rehearsal, corrective feedback, and positive reinforcement to facilitate learning. In the modified version of CBSST used in this project: 1) we will strengthen the focus on corrective feedback from successful social interactions; 2) focus on normalization and destigmatization of attenuated psychotic symptoms; 3) add motivational interviewing techniques to promote treatment engagement; and 4) use examples and role plays. CBSST will be delivered in three 6-session modules (i.e., Cognitive Skills, Social Skills, and Problem Solving Skills), a total of 18 90-minute group sessions.
  Interventions: Behavioral: Cognitive behavioral social skills
- Psychoeducation (Active Comparator): The purpose of this alternative treatment is to match CBSST for the nonspecific effects of therapist contact and interest, social interaction and support. Common factors include client expectancy, providing a rationale for change, therapist factors and therapeutic alliance. The psychoeducation group will meet weekly, for a total of 18 90-minute sessions. Therapists will follow brief guidelines as to what they can and cannot do. In each session the therapists will ask how the previous week had been. Any crises will be dealt with, and advice will be offered to help with any immediate problems. No active CBT or SST techniques will be taught or used. Psychoeducational information about high risk for psychosis will be offered. There will be a focus on listening, reflecting and empathizing, and demonstrating uncritical acceptance and genuineness. Social exchanges amongst participants will be encouraged.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive behavioral social skills
  Arms: Cognitive behavioral social skills
Behavioral: Psychoeducation
  Arms: Psychoeducation

SUMMARY:
Schizophrenia and other psychotic disorders are serious and debilitating mental illnesses that incur substantial suffering for patients and major challenges to the investigators health care and legal systems. The prodrome is the period prior to onset of psychosis when functional decline and clinical symptoms gradually emerge. The presence of a clinical high-risk (CHR) syndrome in young adults is associated with heightened risk (25-35%) for the later development of psychosis, and for those who do not necessarily go on to develop a psychotic illness, research has suggested that the majority continue to have fluctuating subthreshold symptoms and poor social and role functioning. There are no specific treatments to help with these functional difficulties. However, recent findings suggest that in people with schizophrenia, Cognitive Behavioral and Social Skills Training (CBSST) leads to significantly greater increase in the frequency of social functioning activities compared to treatment as usual or goal-focused supportive therapy, and preliminary data suggest CBSST is a feasible treatment for CHR. This proposal is a competitive application for a three-site, longitudinal study aimed at testing the effectiveness and feasibility as well as mediators and mechanisms of action of a manualized CBSST intervention that will target functional difficulties associated with clinical risk states for psychosis. The goals are 1) to examine whether CBSST compared to a placebo intervention (psychoeducation) matched for group involvement and therapist time improves functioning in youth at CHR and 2) to determine whether reduction in defeatist beliefs and improvement in social competence mediate change in psychosocial functioning in CHR youth in the CBSST. In this single-blind randomized 2-arm trial participants will be randomized to one of two treatments: CBSST, an 18-week group comprised of three modules; 1) Cognitive Skills; 2) Social Skills; and 3) Problem Solving, or a psychoeducation support group that does not teach active cognitive behavioral therapy or social skills training. Over a five-year period, the multi-site collaboration will follow large CHR sample that will undergo comprehensive assessments of psychosocial and behavioral changes, to examine changes in social and role functioning, as well as symptom changes from baseline to the end of treatment, and to 6 month follow-up. This approach will demonstrate the feasibility of a treatment for which it is easy to train therapists and which can readily be disseminated to regular clinical community practice. In addition, it will provide insights into likely approaches to halting or mitigating the pathological process and advance the investigators understanding of risk prediction; both critical steps in prevention.

ELIGIBILITY:
Inclusion Criteria:

* have prodromal criteria in the past 4 years
* one attenuated psychotic symptom rated 3 or more
* rating on social functioning <6

Exclusion Criteria:

* meet criteria for a psychotic disorder neurological disorder IQ<70

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 203 (Actual)
Dates: Start 2015-01; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Change in the Global Social Functioning Scale | 6 and 12 months
  This is a clinical rating scale that will be given to all participants at baseline, then 6 months which is the end of treatment and then 6 months after the end of treatment so approximately 12 months after baseline to determine if there is an improvement in social functioning

SECONDARY OUTCOMES:
Change in Defeatist Beliefs | 6 and 12 months
  This is a clinical rating scale that will be administer at the end of treatment (6 months) and 6 months after the end of treatment (12 months). This will be administered to all participants

CONTACTS AND LOCATIONS:
Overall Officials: Jean M Addington, PhD, Principal Investigator — University of Calgary
Locations (1):
- Mathison Centre for Research and Education, University of Calgary, Calgary, Alberta, Canada